CLINICAL TRIAL: NCT03661892
Title: Title A Pilot Trial to Evaluate Syndros in Decreasing Opioid Requirement in Patients With Bone Metastases From Breast Cancer
Brief Title: Pilot, Syndros, Decreasing Use of Opioids in Breast Cancer Subjects With Bone Mets
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1808852902; NCI-2018-01916 (Registry Identifier: NCI Trial Identifier)
Record Dates: First submitted 2018-09-05; First posted 2018-09-07 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Bone Metastases; Breast Cancer; Pain
Keywords: Breast Cancer; Bone Metastases; Pain; Opioid; Syndros; Bone pain
MeSH Terms: conditions — Breast Neoplasms; Pain | interventions — Dronabinol

STUDY DESIGN:
Intervention Model Description: This a prospective single arm study enrolling patients (n=20) with bone metastases form breast cancer who have been on opioid therapy for bone pain for at least 4 weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (Syndros) (Experimental): All patients start on Syndros at 4.2 mg po BID for 3 days, if tolerated without side effects the dose is increased to 8.4 mg QAM and 4.2 mg QPM for an additional 3 days. If the patient continues to tolerate the medication, the dose will be increased to 8.4 mg BID for the rest of the study period (total of 8wks).
  Interventions: Drug: Syndros

INTERVENTIONS:
Drug: Syndros — As noted in arm description. For patients who have side effects secondary to Sydnros, the dose will be decreased as below:
  Dose subject is taking Reduction recommendation 8.4mg BID Decreased to 8.4mg AM , 4.2mg PM (or it can be 4.2g in AM and 8.4mg in PM- depending on their side effect timing) 8.4mg AM, 4.2mg PM (or vice versa) 4.2mg BID 4.2mg BID 4.2mg once a day 4.2mg once a day Stop and take off study
  Other Names: Dronabinol

SUMMARY:
In patients with cancer induced bone pain, addition of Syndros will improve pain relief and decrease opioid requirement.

DETAILED DESCRIPTION:
This a prospective single arm study enrolling patients with bone metastases from breast cancer who have been on opioid therapy for bone pain for at least 4 weeks. All patients start on Syndros at 4.2 mg po BID for 3 days, if tolerated without side effects the dose is increased to 8.4 mg QAM and 4.2 mg QPM for an additional 3 days. If the patient continues to tolerate the medication, the dose will be increased to 8.4 mg BID for the rest of the study period (total of 8wks). For patients who have side effects secondary to Sydnros, the dose will be decreased. Side effect assessment will be done by the research team 2 days after making the dose adjustment. If subject continues to have side effects, dose will be held until resolution of symptoms. If the study medicine is held for more than a week continuously, they will be taken off the study. In addition, they will have baseline blood and urine collected for biomarkers and also complete study related questionnaires (for secondary end points). They are also provided an opioid drug diary which they will take home during visit 1 to record their opioid pain medication use. Research staff will be calling patients on a weekly basis to reinforce opioid drug diary, assess for Syndros side effect, and adjust dose of Syndros. At the end of 8 weeks blood and urine is collected again and they will complete the study questionnaires.

ELIGIBILITY:
Inclusion Criteria:

1. Be capable of understanding the investigational nature of the study and all pertinent aspects of the study
2. Be capable of signing and providing written consent in accordance with institutional and federal guidelines
3. Have metastatic breast cancer with bone metastases
4. Be willing and able to comply with scheduled visits, treatment plan, and follow up with research staff
5. Age ≥ 21 years
6. Must be on opioid therapy for bone pain for at least 4 weeks

Exclusion Criteria:

1. Have a known sensitivity to dronabinol or alcohol
2. Have a history of hypersensitivity reaction to alcohol
3. Using medical marijuana currently
4. Using Syndros for nausea or appetite stimulant
5. Receiving or have received disulfiram- or metronidazole- containing products within past 14 days
6. Are currently pregnant or are of child-bearing age and refuse to use adequate contraception
7. Have a history of psychiatric illness
8. Have a history of seizure disorders

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-12-19 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2021-04-26 (Actual)

PRIMARY OUTCOMES:
Need for opiate pain medication | Eight weeks
  To evaluate change in opiate pain medication use after addition of Syndros.Hypothesis: Syndros will decrease the opiate usage by at least 20% at the end of 8wks. We will evaluate opioid pain medication use by using a drug diary and assessing the percentage change in opiate pain medication requirement at end of 8wks.

SECONDARY OUTCOMES:
Change in pain | Eight weeks
  To evaluate change in pain using the Brief Pain Inventory tool. Hypothesis: Addition of Syndros will decrease pain intensity on the rating tool.
Change in quality of life | Eight weeks
  2. To evaluate change in quality of life using the EORTC QLQ-C30 version 3.0 questionnaire. Hypothesis: Addition of Syndros will improve quality of life.
Change in bone modulation | Eight weeks
  To evaluate change in bone modulation by Syndros. Hypothesis: Syndros will decrease bone degradation there by decreasing serum and urine C-terminal telopeptide collagen cross-linker (CTX), N-terminal telopeptide (NTX) and increase osteocalcin.

CONTACTS AND LOCATIONS:
Overall Officials: Pavani Chalasani, MD, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No